CLINICAL TRIAL: NCT03553212
Title: Twice High Dose External Beam Radiotherapy by Image-guided Tomotherapy for Organ-confined Prostate Cancer Treatment Emulating HDR Brachytherapy: Single Institution Feasibility Study
Brief Title: Twice High Dose External Beam Radiotherapy by Image-guided Tomotherapy for Organ-confined Prostate Cancer Treatment Emulating High Dose Radiation (HDR) Brachytherapy
Acronym: THRIP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: outdated, progress in clinical practice.
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST185.06
Record Dates: First submitted 2018-05-16; First posted 2018-06-12 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Prostate Adenocarcinoma; Radiotherapy; Complications; Tomotherapy
Keywords: Prostate cancer; organ-confined; external beam Radiotherapy; Image-guided tomotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Intervention Model Description: Feasibility trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High dose external beam Radiotherapy (Experimental): Image-guided tomotherapy
  Interventions: Radiation: tomotherapy

INTERVENTIONS:
Radiation: tomotherapy — 20-23 Gy in 2 fractions on the whole prostate gland +/- seminal vesicles and 24-27 Gy in 2 fractions as simultaneous integrated boost (SIB) on the dominant intraprostatic lesion (DIL) 2 weeks in all.

SUMMARY:
Feasibility trial of twice high dose radiotherapy using Tomotherapy in patients with organ confined Prostate Cancer histologically proven. The study involves 2 steps:

A) Assessment of safety as proportion of patients with acute ≥G3 Genito-urinary (GU) and Gastro-intestinal (GI) side effects on the first 16 enrolled patients; B) evaluation of primary and secondary objectives on overall patients.

DETAILED DESCRIPTION:
Twice High dose external beam Radiotherapy by Image-guided tomotherapy for organ-confined Prostate cancer treatment emulating HDR brachytherapy:

Feasibility trial of twice high dose radiotherapy using Tomotherapy in patients with organ confined Prostate Cancer histologically proven. The study involves 2 steps:

A) Assessment of safety as proportion of patients with acute ≥G3 Genito-urinary (GU) and Gastro-intestinal (GI) side effects on the first 16 enrolled patients; B) evaluation of primary and secondary objectives on overall patients. Thirty-one patients will be enrolled, with histologically confirmed very low , low and intermediate risk prostate cancer following the National Comprehensive Cancer Network (NCCN) risk categories guidelines. Patient should not be eligible to prostatectomy or patient's should refuse to undergo surgery.

Prescription dose to the target: 20-23 Gy in 2 fractions on the whole prostate gland +/- seminal vesicles and 24-27 Gy in 2 fractions as simultaneous integrated boost (SIB) on the dominant intraprostatic lesion (DIL) 2 weeks in all.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma (a diagnostic biopsy with at least 10 cores is needed)
* Low and intermediate-risk NCCN risk categories: low-risk ( cT1-2a, Gleason Score ≤ 6 PSA <10 ng/ml) and among those with intermediate-risk features (clinical stage T2b-c or GS 7 or PSA 10-20 ng/ml) those patients with favorable ones (a single factor for intermediate risk and GLS 3 + 4 and <50% of biopsy cores containing cancer) will be selected. (30).
* Age ≥18 years
* Good performance status , Eastern Cooperative Oncology Group (ECOG) < 2) or Karnofsky performance status (KPS) > 70
* No previous pelvic RT
* Patient not eligible to prostatectomy or patient's refusal to undergo surgery.
* NO previous prostatectomy or TURP
* Good urinary flow (peak flow ≥ 10 ml/s)
* Previous ADT is permitted
* Prostate size ≤ 60 cc
* International Prostate Symptom Score ≤ 15
* Male participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 3 months thereafter
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Nodal involvement or distant metastases (cN1 or cM1)
* Extracapsular tumor or locally advanced disease (cT3-cT4)
* IPSS questionnaire > 20
* Concomitant inflammatory bowel
* Prior history of chronic prostatitis
* Prior history of urethral stricture
* Important systemic diseases or oral anticoagulant therapy ongoing
* Non-conformity to dose constraints at the treatment planning
* Other invasive cancer (apart from non-melanoma skin), unless the patient has been free from disease for at least 3 years;
* Abnormal complete blood count. Any of the following: platelet count less than 75,000/ml, Hb level less than 10 gm/dl, WBC less than 3.5/ml, abnormal renal function tests (creatinine > 1.5), severe renal impairment (GFR less than 30)
* Placement of pacemakers and metallic vascular clips (all contraindication to performing prostate mpMRI).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
occurrence of Grade ≥3 early GU toxicity | within 3 months after end of Radiotherapy
  Early Grade ≥3 GU toxicity measured by Radiation Therapy Oncology Group and European Organisation for Research and Treatment of Cancer (RTOG/EORTC) toxicity scale, using a scoring range from 0 to 5 for, where 0 means an absence of radiation effects and 5 means the effects led to death
occurrence of Grade ≥3 early GI toxicity | within 3 months after end of Radiotherapy
  Early Grade ≥3 GI toxicity measured by Radiation Therapy Oncology Group and European Organisation for Research and Treatment of Cancer (RTOG/EORTC) toxicity scale, using a scoring range from 0 to 5 for, where 0 means an absence of radiation effects and 5 means the effects led to death

SECONDARY OUTCOMES:
Occurrence of Grade ≥3 Late GU toxicity | more than 6 months after end of Radiotherapy
  Late Grade ≥3 GU toxicity measured by Radiation Therapy Oncology Group and European Organisation for Research and Treatment of Cancer (RTOG/EORTC) toxicity scale, using a scoring range from 0 to 5 for, where 0 means an absence of radiation effects and 5 means the effects led to death
Evaluation of Prostate Antigen Serum (PSA) failure | up to 8 years
  Evaluation of PSA failure is defined according to the Consensus Statement of the American Society of Radiation Oncology (ASTRO) as elevation of PSA levels nadir +2 ng/ml and confirmed by one measurement (Phoenix criterion) or biochemical response through trimestral PSA level evaluation.
Time to biochemical failure (TTBF) | up to 8 years
  the time frame from the beginning date of radiation therapy (RT) to the date of PSA failure;
Time to progression (TTP) | up to 8 years
  time to progression (TTP), both local and distant defined as time from beginning date of RT to the date of progression of disease, both local and distant, or death whichever came first;
Overall Survival (OS) | up to 8 years
  overall survival, defined as the time from the start of treatment to the date of death from any cause, if data will be available, also cause specific survival will be calculated.
Quality of Life (QoL) | before treatment, at 12 and 24 months of follow up
  Treatment-related quality of life (QoL) according to the Functional Assessment of Cancer Therapy (FACT-Prostate) questionnaire; which consists of 39 items. Each item is rated on a 0 to 4 Likert type scale, and then combined to produce subscale scores. Higher scores represent better QoL.
Quality of urinary function | before treatment, at 3, 6, 12 and 24 months of follow up
  Urinary functions according to the International Prostate symptom Score (IPSS) questionnaire, which consists of 7 items. Each item is rated on a 0 to 5 score to produce a total I-PSS score with a range from 0 to 35 (asymptomatic to very symptomatic).
Quality of erectile function | before treatment, at 3, 6, 12 and 24 months of follow up
  Erectile functions according to International Index of Erectile Function (IEEF-5) questionnaire, which consists of 5 items. Each item is rated on a 1 to 5. High scores represent better erectile function.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Pia Colangione, MD, Study Chair — Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST)
Locations (1):
- Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola, FC, Italy